CLINICAL TRIAL: NCT07258810
Title: Evaluation of Tolerance and Quality of Life in Patients With Neuroendocrine Tumors Treated With Oral Anti-Tumor Drugs Within a Therapeutic Education Program
Acronym: ETP-NET
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0703; 2025-A01985-44 (Other: ID-RCB)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine (NE) Tumors; Oral Anti-Tumor Drugs; Therapeutic Education Program
Keywords: Neuroendocrine tumor; Oral Anti-Tumor Drugs; Therapeutic Education Program; Tolerance; Quality of Life
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients enrolled in the therapeutic education program: Patient with a neuroendocrine tumor requiring treatment with oral antitumor therapy
  Interventions: Other: Questionnaires
- Patients not enrolled in the therapeutic education program: Patient with a neuroendocrine tumor requiring treatment with oral antitumor therapy
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — questionnaires given to patients in both groups: treatment adherence (MMAS-4 scale) at months 1 and 3, quality of life (EORTC QLQ-C30) at months 0, 1 and 3, and a satisfaction questionnaire developed and validated by the healthcare team and members of the French patient association for individuals with various neuroendocrine tumors (APTED) at month 3.

SUMMARY:
In recent years, the arrival of targeted oral therapies has greatly changed cancer treatment. These therapies help patients stay independent by reducing the number of hospital visits, since the treatment is given at home. However, this way of giving treatment brings specific challenges, especially in managing side effects and making sure patients follow their treatment properly.

Because of this, many patient education programs have been created to help patients learn how to manage their treatment on their own. Although only a few studies have formally looked at how useful these programs are, the available information suggests that they help patients handle side effects better and follow their treatment more closely.

Neuroendocrine tumors are a diverse group of tumors that are becoming more common. More patients with these tumors are now treated with targeted oral therapies such as everolimus, sunitinib, cabozantinib, or chemotherapy with temozolomide and capecitabine.

These treatments are often given together with a patient education program. However, so far, no study has specifically looked at how helpful these education programs are for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years) at the time of the study
* Patient diagnosed with a neuroendocrine tumor (NET) with an indication for treatment with oral anti-tumor agents (everolimus, sunitinib, cabozantinib, temozolomide +/- capecitabine, others including lenvatinib)
* Collection of the patient's non-opposition to participate in the study

Exclusion Criteria:

* Minors
* Pregnant, parturient, or breastfeeding women
* Persons deprived of liberty by judicial or administrative decision
* Adults under legal protection measures (guardianship, conservatorship)
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will be carried out among patients hospitalized in the Medical Oncology department at Edouard Herriot University Hospital.
  Every consecutive patient with an indication for oral anti-tumor agents (ATO) within the context of a neuroendocrine tumor (NET) will be screened and included in the study in the absence of contraindications and after obtaining their non-opposition.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the incidence of grade 3 to 5 adverse events in patients with neuroendocrine tumors treated with oral anti-tumor agents (ATO), based on their participation in a therapeutic education program | at 3 months
  * Adverse effects (CTCAE v5.0) within 3 months following the initiation of ATO Grade 3-4 and 5 adverse effects: hematological, digestive, cutaneous, renal, hepatic toxicity (cytolysis >5x normal), cardiovascular (including arterial hypertension and thromboembolic complications), pulmonary (interstitial lung disease), metabolic (including hyperglycemia, lipid profile abnormalities)
  * Actions taken at Month 1 and Month 3 Treatment suspension or delay of the cycle: number of suspensions, duration of suspension (in days) or number of cycle delays, duration of delay (in days) Dose reduction: reduction (yes/no), new dose Hospitalization due to adverse effects: number of hospitalizations, duration (total number of hospitalization days)
  * Description of patient follow-up and therapeutic patient education program Number of consultations: teleconsultation or in-person consultation, with nurse or physician (general practitioner or oncologist) Number of phone calls: with nurse or physician

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gerard, Dr, Principal Investigator — Medical Oncology Department
Locations (1):
- Edouard Herriot University Hospital, Lyon, France